CLINICAL TRIAL: NCT02206750
Title: The Interaction of Social Factors With Air Pollution
Acronym: SOZIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Diaz-Sanchez, Chief, Clinical Research Branch, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: # 13-1644
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Exposure to Environmental Pollution, Non-occupational
Keywords: Controlled Human exposure study; Air Pollution; Cardiovascular; Social factors; Cognitive function
MeSH Terms: interventions — Environment, Controlled; Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clean Air (Sham Comparator): Exposure to clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: Clean Air
- Ozone (Experimental): Exposure to ozone will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus.
  Interventions: Other: Ozone

INTERVENTIONS:
Other: Clean Air — Each subject will be exposed to clean air for 2 hours. Subjects will exercise on a bike or treadmill. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/min/m2BSA followed by a 15 minute rest period.
  Arms: Clean Air
Other: Ozone — Each subject will be exposed up to 0.3ppm ozone for 2 hours. Subjects will exercise on a bike or treadmill. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/min/m2BSA followed by a 15 minute rest period.
  Other Names: O3
  Arms: Ozone

SUMMARY:
Purpose:

The purpose of this protocol is to understand how social factors such as psychosocial stress may modify how people respond to air pollution. Ultimately this will help us understand health disparities from poor air quality.

Participants:

Up to 40 healthy adults,18-33 years old with different perception of stress will participate and complete this study.

Procedures (methods):

Subjects will be exposed to clean air and to ozone ( 300ppb) for 2 hours in a controlled environment chamber. Cardiac, vascular, pulmonary and cognitive function will be evaluated pre, immediately post and 18 hr post exposure.

The primary endpoint will be Heart Rate Variability . Secondary endpoints will include pulmonary function, analysis of blood clotting/coagulation factors, biomarkers of stress, cognitive function, radial artery pulse wave measurements and analysis of soluble factors present in plasma.

DETAILED DESCRIPTION:
Over the past decades, air quality in the U.S. has improved significantly. Even so, millions of people in the U.S. still live in counties that do not meet air quality standards for one or more pollutants. Ozone is a major component of photochemical smog and is one of the most thoroughly studied gaseous pollutants. Controlled human exposure studies have been critical in demonstrating that it can cause airway inflammation 1-3, including increases in neutrophil infiltration into the lung and the production of pro-inflammatory mediators 4,5[, and ultimately decrements in lung function [reviewed in 6]. More recent studies have shown that ozone can also increase vascular inflammation, as well as alter autonomic nervous system control of heart rate and cardiac repolarization 7. Numerous epidemiological studies have also demonstrated an association between acute and chronic exposure to ambient levels of ozone and various health effects most notably asthma 6. These studies have also highlighted a need to incorporate social and nonchemical factors into risk assessments 8. Similarly, social factors such as psychological stress are now regarded as important contributors to asthma outcomes 9,10. This protocol is aimed at investigating how stress impacts health responses to air pollutants. Since psychosocial stress-related susceptibility has been proposed to explain social disparities, this will help us understand which populations and individuals are at increased risk from air pollution.

This protocol is designed to determine whether nonchemical stressors exacerbate ozone effects. In particular we will focus on elevated psychosocial stress as it has been shown to contribute to several adverse health outcomes, most notably, to cardiovascular disease. The physiological mechanism by which psychosocial stress leads to health effects is due, at least in part, to elevated circulating glucocorticoids, or stress hormones, which are regulated by the hypothalamic-pituitary-adrenal (HPA). In the last 30 years the concept of allostasis has evolved. Allostasis is the process whereby an organism adapts to the demands of the environment. An allostatic load model applies this concept to chronic stress11. In this model the perception of threat over long time intervals (perceived stress) can cause over-activation of the HPA-axis resulting in changes in physiological systems as chemical imbalances in autonomic nervous system, central nervous system, neuroendocrine, and immune system activity. Factors such as genetics, behavior, life events and diet can impact this model. To our knowledge no clinical study has investigated the link between air pollution effects on cardiovascular disease and psychosocial stress. However, several studies have now shown an association between stress and respiratory outcomes to air pollution. Claugherty and colleagues (2007) found an association between traffic-related air pollution and asthma solely among children exposed to violence 12. Shankardass and colleagues demonstrated that children from stressful households are more susceptible to the effects of traffic-related pollution on the development of asthma 13. In that study, stress was evaluated using the Perceived Stress Scale (PSS) developed by Dr. Sheldon Cohen of Carnegie Mellon University. This is the most widely used psychological instrument for measuring the perception of stress and has been validated in multiple studies. We will use this scale to evaluate the degree to which subjects appraise situations in their life as stressful. Heart rate variability (HRV) is considered to be a reliable biomarker of stress. Chronic stress has been shown to be associated with decreases in HRV 14. Since acute ozone exposure can also cause changes in HRV, we have chosen HRV as our primary endpoint. We hypothesize that the imbalance between the sympathetic and the parasympathetic nervous system caused by chronic stress will result in altered responses to ozone exposure that will be reflected by HRV.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 and 33 years of age.

  1. 4-point Perceived Stress Symptom score <2 or >6
  2. Physical conditioning allowing intermittent, moderate exercise for two hours.
  3. Ability to complete the exposure exercise regimen without reaching 80% of predicted maximal heart rate.

     Predicted maximal heart rate will be calculated using the equation (described by Tanaka et al. [2001] J. Am. Coll. Cardiol.): [208bpm-((0.7) x (age in years))]
  4. Normal baseline 12-lead resting EKG, or if the automated reading is not normal the EKG must be approved by a study cardiologist.
  5. Normal lung function Forced vital capacity (FVC) ≥ 80% of that predicted for gender, ethnicity, age and height (according to NHANESIII guidelines).

     Forced expiratory volume in one second (FEV1) ≥ 80%of that predicted for gender, ethnicity, age and height.

     FEV1/FVC ratio ≥ 80% of predicted values.
  6. Oxygen saturation ≥ 96% on room air.

Exclusion Criteria:

* . Individuals with a history of acute or chronic cardiovascular disease, chronic respiratory disease, diabetes, rheumatologic diseases, or immunodeficiency state.

  2. Individuals with a Framingham risk score (Hard Coronary Heart Disease; HCHD; 10-year risk) ≥10.

  3. Individuals with asthma or a history of asthma. 4. Individuals who are allergic to chemical vapors or gases. 5. Females who are pregnant, attempting to become pregnant, or breastfeeding. 6. Individuals that are unwilling or unable to stop taking vitamin C or E, or medications that may impact the results of ozone challenge such at least two weeks prior to the study and for the duration of the study. Medications not specifically mentioned here may be reviewed by the investigators prior to an individual's inclusion in the study.

  7. Individuals who have smoked tobacco during the last five years or those with a history of >5 pack years.

  8. Individuals living with a smoker who smokes inside the house. 9. Individuals with a body mass index (BMI) >35 or <18. Body mass index is calculated by dividing the weight in kilograms by the square of the height in meters.

  10. Individuals with occupational exposures to high levels of vapors, dust, gases, or fumes on an on-going basis.

  11. Individuals with uncontrolled hypertension (≥150 systolic or ≥90 diastolic).

  12. Individuals that do not understand or speak English. 13. Individuals that are unable to perform the exercise required for the study. 14. Individuals that are taking beta blocker medications. 15. Individuals with a history of skin allergies to adhesives used in securing EKG electrodes.

  16. Individuals with unspecified diseases, conditions, or medications that might influence the responses to the exposures, as judged by the medical staff.

  17. Individuals that are unwilling or unable to stop taking over-the-counter pain medications such as aspirin, ibuprofen (Advil, Motrin), naproxen (Aleve), or other non-steroidal anti-inflammatory ("NSAID") medications for 48 hours prior to the exposures and post-exposure visits.

  18. Individuals that are taking systemic steroids or beta-blocker medications. 19. Individuals with a hemoglobin A1c (HbA1c) level > 6.4%.

Temporary Exclusion Criteria

1. Individuals with active seasonal allergies during the time of participation in the study.
2. Individuals suffering from acute respiratory illness within four weeks prior to any of the study exposure series.
3. Individuals that have been exposed to smoke and fumes within 24 hours of any study visit.
4. Individuals that have consumed alcohol within 24 hours of any study visit.
5. Individuals that have engaged in strenuous exercise within 24 hours of any study visit.
6. Individuals that have been exposed to ozone-based home air purifiers within 24 hours of any study visit.
7. Individuals that have been exposed to unvented household combustion sources (gas stoves, lit fireplaces, oil/kerosene heaters) within 48 hours of any study visit.

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability | Pre exposure to 24hours post exposure
  10 minute electrocardiogram recording (measured by Holter ECG) in which the subject has been resting for 20 minutes prior. Collected on a Mortara H12+ 12-Lead ECG Recorder (Mortara Instrument, Inc., Milwaukee, WI). The digitally recorded ECGs are sampled at 180 Hz.

SECONDARY OUTCOMES:
Forced expired volume in the first second (FEV1) | Pre exposure to 24hours post exposure
  Forced expired volume in the first second (FEV1) is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Index of clotting/coagulation factor | Pre exposure to 24hours post exposure
  Index of clotting/coagulation factors are the mean % changes in a basket of clotting/coagulation factors (d-dimer, PA-1, tPA, vWillebrand factor and plasminogen) in the blood following exposure to ozone vs. clean air.
Forced Vital Capacity | Pre exposure to 24hours post exposure
  Forced Vital Capacity(FVC) is determined by spirometry performed on a dry seal spirometer interfaced to a computer.
Index of inflammatory markers | Pre exposure to 24hours post exposure
  Index of inflammatory markers is the mean % changes in a basket of factors related to systemic inflammation (IL-6, IL-8, TNF-a, IL-b, CRP) in the blood following exposure to ozone vs. clean air.
Cortisol | Pre exposure to 24hours post exposure
  The mean % change of cortisol levels in the blood following exposure to ozone vs. clean air.
Cognitive function performance | Pre exposure to 24hours post exposure
  Index of cognitive function tests measured using six tests of the Cantab Research Suite (Reaction Time Test (RTI), Attention Switching Task (AST), Spatial Working Memory (SWM), Paired Associate Learning (PAL), Rapid Visual Information Processing (RVP), and Stop Signal Task (SST)) following exposure to ozone vs. clean air.

CONTACTS AND LOCATIONS:
Overall Officials: David Diaz-Sanchez, PhD, Principal Investigator — U.S. Environmental Protection Agency
Locations (1):
- U.S. EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Devlin RB, McDonnell WF, Becker S, Madden MC, McGee MP, Perez R, Hatch G, House DE, Koren HS. Time-dependent changes of inflammatory mediators in the lungs of humans exposed to 0.4 ppm ozone for 2 hr: a comparison of mediators found in bronchoalveolar lavage fluid 1 and 18 hr after exposure. Toxicol Appl Pharmacol. 1996 May;138(1):176-85. doi: 10.1006/taap.1996.0111. PMID 8658507
- [Background] Devlin RB, McDonnell WF, Mann R, Becker S, House DE, Schreinemachers D, Koren HS. Exposure of humans to ambient levels of ozone for 6.6 hours causes cellular and biochemical changes in the lung. Am J Respir Cell Mol Biol. 1991 Jan;4(1):72-81. doi: 10.1165/ajrcmb/4.1.72. PMID 1846079
- [Background] Schelegle ES, Siefkin AD, McDonald RJ. Time course of ozone-induced neutrophilia in normal humans. Am Rev Respir Dis. 1991 Jun;143(6):1353-8. doi: 10.1164/ajrccm/143.6.1353. PMID 2048824
- [Background] Bascom R, Naclerio RM, Fitzgerald TK, Kagey-Sobotka A, Proud D. Effect of ozone inhalation on the response to nasal challenge with antigen of allergic subjects. Am Rev Respir Dis. 1990 Sep;142(3):594-601. doi: 10.1164/ajrccm/142.3.594. PMID 2202248
- [Background] Peden DB, Setzer RW Jr, Devlin RB. Ozone exposure has both a priming effect on allergen-induced responses and an intrinsic inflammatory action in the nasal airways of perennially allergic asthmatics. Am J Respir Crit Care Med. 1995 May;151(5):1336-45. doi: 10.1164/ajrccm.151.5.7735583.
- [Background] Devlin RB, Duncan KE, Jardim M, Schmitt MT, Rappold AG, Diaz-Sanchez D. Controlled exposure of healthy young volunteers to ozone causes cardiovascular effects. Circulation. 2012 Jul 3;126(1):104-11. doi: 10.1161/CIRCULATIONAHA.112.094359. Epub 2012 Jun 25. PMID 22732313
- [Background] Gray SC, Edwards SE, Schultz BD, Miranda ML. Assessing the impact of race, social factors and air pollution on birth outcomes: a population-based study. Environ Health. 2014 Jan 29;13(1):4. doi: 10.1186/1476-069X-13-4. PMID 24476365
- [Background] Wright RJ. Epidemiology of stress and asthma: from constricting communities and fragile families to epigenetics. Immunol Allergy Clin North Am. 2011 Feb;31(1):19-39. doi: 10.1016/j.iac.2010.09.011. PMID 21094921
- [Background] Wright RJ, Schreier HM. Seeking an integrated approach to assessing stress mechanisms related to asthma: is the allostatic load framework useful? Am J Respir Crit Care Med. 2013 Jan 15;187(2):115-6. doi: 10.1164/rccm.201210-1816ED. No abstract available. PMID 23322789
- [Background] Juster RP, McEwen BS, Lupien SJ. Allostatic load biomarkers of chronic stress and impact on health and cognition. Neurosci Biobehav Rev. 2010 Sep;35(1):2-16. doi: 10.1016/j.neubiorev.2009.10.002. Epub 2009 Oct 12. PMID 19822172
- [Background] Clougherty JE, Levy JI, Kubzansky LD, Ryan PB, Suglia SF, Canner MJ, Wright RJ. Synergistic effects of traffic-related air pollution and exposure to violence on urban asthma etiology. Environ Health Perspect. 2007 Aug;115(8):1140-6. doi: 10.1289/ehp.9863. PMID 17687439
- [Background] Shankardass K, McConnell R, Jerrett M, Milam J, Richardson J, Berhane K. Parental stress increases the effect of traffic-related air pollution on childhood asthma incidence. Proc Natl Acad Sci U S A. 2009 Jul 28;106(30):12406-11. doi: 10.1073/pnas.0812910106. Epub 2009 Jul 20. PMID 19620729
- [Background] Schubert C, Lambertz M, Nelesen RA, Bardwell W, Choi JB, Dimsdale JE. Effects of stress on heart rate complexity--a comparison between short-term and chronic stress. Biol Psychol. 2009 Mar;80(3):325-32. doi: 10.1016/j.biopsycho.2008.11.005. Epub 2008 Dec 3. PMID 19100813